CLINICAL TRIAL: NCT03983954
Title: Phase 1B, Open-Label, Dose Escalation and Cohort Expansions Trial of Naptumomab Estafenatox (NAP, ABR-217620) in Combination With Durvalumab (MEDI4736) in Subjects With Selected Advanced or Metastatic Solid Tumors
Brief Title: Naptumomab Estafenatox in Combination With Durvalumab in Subjects With Selected Advanced or Metastatic Solid Tumor, Including a Cohort Expansion in Esophageal Cancer.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NeoTX Therapeutics Ltd. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 127-CL-01 (NT-NAP-101)
Record Dates: First submitted 2019-05-27; First posted 2019-06-12 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: ER+ Breast Cancer; Ovarian Cancer; Cervical Squamous Cell Carcinoma; Pancreatic Adenocarcinoma; Endometrial Cancer; Renal Cell Carcinoma; Urothelial Cancer; Head and Neck Squamous Cell Carcinoma; Mesothelioma; Melanoma; Hepatocellular Carcinoma; Prostate Cancer; NSCLC; HER2-negative Breast Cancer; Triple Negative Breast Cancer; Bladder Cancer; Colorectal Cancer Metastatic; GastroEsophageal Cancer; NSCL2 Gene Mutation; Esophageal Cancer
Keywords: Esophageal cancer; Squamous cell carcinoma of the esophagus; Adenocarcinoma of the esophagus
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Carcinoma, Renal Cell; Squamous Cell Carcinoma of Head and Neck; Mesothelioma; Melanoma; Carcinoma, Hepatocellular; Prostatic Neoplasms; Triple Negative Breast Neoplasms; Urinary Bladder Neoplasms; Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — obinutuzumab; naptumomab estafenatox; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Dose Escalation naptumomab estafenatox 2 µg/kg and durvalumab (Experimental): NAP was administered on the first four days of each 21-day cycle, at daily doses of 2 µg/kg. Durvalumab (1120 mg, IV, 1- 1.5 hours after completion of the administration of NAP) was administered on the second day of each 21-day cycle. After cycle 3, patients continued to receive durvalumab alone at a dose of 1500 mg delivered once every 28 days, until confirmed disease progression or unacceptable toxicity for a maximum of up to 24 months.
  Interventions: Combination Product: Naptumomab estafenatox and durvalumab
- Dose Escalation naptumomab estafenatox 5 µg/kg and durvalumab (Experimental): NAP was administered on the first four days of each 21-day cycle, at daily doses of 5 µg/kg. Durvalumab (1120 mg, IV, 1- 1.5 hours after completion of the administration of NAP) was administered on the second day of each 21-day cycle. After cycle 3, patients continued to receive durvalumab alone at a dose of 1500 mg delivered once every 28 days, until confirmed disease progression or unacceptable toxicity for a maximum of up to 24 months.
  Interventions: Combination Product: Naptumomab estafenatox and durvalumab
- Dose Escalation naptumomab estafenatox 10 µg/kg and durvalumab (Experimental): NAP was administered on the first four days of each 21-day cycle, at daily doses of 10 µg/kg. Durvalumab (1120 mg, IV, 1- 1.5 hours after completion of the administration of NAP) was administered on the second day of each 21-day cycle. After cycle 3, patients continued to receive durvalumab alone at a dose of 1500 mg delivered once every 28 days, until confirmed disease progression or unacceptable toxicity for a maximum of up to 24 months.
  Interventions: Combination Product: Naptumomab estafenatox and durvalumab
- Dose Escalation naptumomab estafenatox 15 µg/kg and durvalumab (Experimental): NAP was administered on the first four days of each 21-day cycle, at daily doses of 15 µg/kg. Durvalumab (1120 mg, IV, 1- 1.5 hours after completion of the administration of NAP) was administered on the second day of each 21-day cycle. After cycle 3, patients continued to receive durvalumab alone at a dose of 1500 mg delivered once every 28 days, until confirmed disease progression or unacceptable toxicity for a maximum of up to 24 months.
  Interventions: Combination Product: Naptumomab estafenatox and durvalumab
- Dose Escalation naptumomab estafenatox 20 µg/kg and durvalumab (Experimental): NAP was administered on the first four days of each 21-day cycle, at daily doses of 20 µg/kg. Durvalumab (1120 mg, IV, 1- 1.5 hours after completion of the administration of NAP) was administered on the second day of each 21-day cycle. After cycle 3, patients continued to receive durvalumab alone at a dose of 1500 mg delivered once every 28 days, until confirmed disease progression or unacceptable toxicity for a maximum of up to 24 months.
  Interventions: Combination Product: Naptumomab estafenatox and durvalumab
- Dose escalation, obinutuzumab pretreatment followed by NAP 10 µg/kg and durvalumab (Experimental): Obinutuzumab (1000 mg/day) was administered on days 13 and 12 prior to the first day of NAP. NAP was administered on the first four days of each 21-day cycle, at daily doses of 10 µg/kg. Durvalumab (1120 mg, IV, 1- 1.5 hours after completion of the administration of NAP) was administered on the second day of each 21-day cycle. After cycle 3, patients continued to receive durvalumab alone at a dose of 1500 mg delivered once every 28 days, until confirmed disease progression or unacceptable toxicity for a maximum of up to 24 months.
  Interventions: Combination Product: Obinutuzumab, naptumomab estafenatox and durvalumab
- Dose escalation, obinutuzumab pretreatment followed by NAP 15 µg/kg and durvalumab (Experimental): Obinutuzumab (1000 mg/day) was administered on days 13 and 12 prior to the first day of NAP. NAP was administered on the first four days of each 21-day cycle, at daily doses of 15 µg/kg. Durvalumab (1120 mg, IV, 1- 1.5 hours after completion of the administration of NAP) was administered on the second day of each 21-day cycle. After cycle 3, patients continued to receive durvalumab alone at a dose of 1500 mg delivered once every 28 days, until confirmed disease progression or unacceptable toxicity for a maximum of up to 24 months.
  Interventions: Combination Product: Obinutuzumab, naptumomab estafenatox and durvalumab
- MTD expansion, obinutuzumab pretreatment with NAP at MTD and durvalumab (Experimental): NAP at 15mcg/kg and durvalumab (1120 mg) were given for 6 cycles after pre-treatment of obinutuzumab (1000 mg/day) on D-13 and D-12. After cycle 6, patients continued to receive durvalumab alone at a dose of 1500 mg delivered once every 28 days, until confirmed disease progression or unacceptable toxicity for a maximum of up to 24 months.
  Interventions: Combination Product: Obinutuzumab, naptumomab estafenatox and durvalumab
- MTD expansion, obinutuzumab pretreatment with NAP, at the previous dose level, and durvalumab (Experimental): NAP, at the previous dose level (10mcg/kg), and durvalumab (1120 mg) were given for 6 cycles after pre-treatment of obinutuzumab (1000 mg/day) on D-13 and D-12. After cycle 6, patients continued to receive durvalumab alone at a dose of 1500 mg delivered once every 28 days, until confirmed disease progression or unacceptable toxicity for a maximum of up to 24 months.
  Interventions: Combination Product: Obinutuzumab, naptumomab estafenatox and durvalumab
- MTD expansion, abbreviated regimen of obinutuzumab pretreatment with NAP at MTD and durvalumab (Experimental): NAP at MTD (10 mcg/kg/day) and durvalumab (1120 mg) were given for 6 cycles after a single dose of pre-treatment of obinutuzumab (1000 mg/day) on D-7. After cycle 6, patients continued to receive durvalumab alone at a dose of 1500 mg delivered once every 28 days, until confirmed disease progression or unacceptable toxicity for a maximum of up to 24 months.
  Interventions: Combination Product: Obinutuzumab, naptumomab estafenatox and durvalumab
- Cohort Expansion in Esophageal Cancer: Obinutuzumab pretreatment, NAP and Durvalumab (Experimental): NAP will be administered at a dose of 10 μg/kg/day by IV bolus on Days 1 through 4 of the first 6 treatment cycles, and durvalumab will be administered at a flat dose of 1120 mg on Day 2 of each of the first 6 treatment cycles. Starting Cycle 7, a single administration of NAP at the same dose and durvalumab at the dose of 1500 mg will be administered on the same day (Day 1) in 28-day treatment cycles. The first 6 treatment cycles will be 21 days in duration and, starting Cycle 7 onward, treatment cycles will be 28 days in duration. Study treatment will continue until disease progression, untoward toxicity, noncompliance, or for a maximum duration of 2 years.
  Interventions: Combination Product: Obinutuzumab, naptumomab estafenatox and durvalumab

INTERVENTIONS:
Combination Product: Obinutuzumab, naptumomab estafenatox and durvalumab — Obinutuzumab is given intravenous (I.V.) 1,000 mg concentrate for solution for infusion, as pre-treatment.
  Dose escalation and MTD Expansion: NAP is given as an intravenous (I.V.) bolus injection at multiple doses.
  Durvalumab is given at a dose of 1120 mg, I.V, 1- 1.5 hours after completion of the administration of NAP on the second day of each 21-day cycle, and when administered as monotherapy at a dose of 1500 mg delivered once every 28 days.
  Esophageal cohort expansion: NAP is given as an intravenous (I.V.) bolus injection at multiple doses on cycles 1-6 and one dose per cycle starting cycle 7. Durvalumab is given at a dose of 1120 mg, I.V, 1- 1.5 hours after completion of the administration of NAP on the second day of each 21-day cycle during cycles 1-6, and at a dose of 1500 mg delivered once every 28 days starting cycle 7.
  Other Names: (ABR-217620; NAP); (IMFINZI; MEDI4736); [Gazyva]
  Arms: Cohort Expansion in Esophageal Cancer: Obinutuzumab pretreatment, NAP and Durvalumab; Dose escalation, obinutuzumab pretreatment followed by NAP 10 µg/kg and durvalumab; Dose escalation, obinutuzumab pretreatment followed by NAP 15 µg/kg and durvalumab; MTD expansion, abbreviated regimen of obinutuzumab pretreatment with NAP at MTD and durvalumab; MTD expansion, obinutuzumab pretreatment with NAP at MTD and durvalumab; MTD expansion, obinutuzumab pretreatment with NAP, at the previous dose level, and durvalumab
Combination Product: Naptumomab estafenatox and durvalumab — NAP was given as an intravenous (I.V.) bolus injection at multiple doses. Durvalumab was given at a dose of 1120 mg, I.V, 1- 1.5 hours after completion of the administration of NAP on the second day of each 21-day cycle, and when administered as monotherapy at a dose of 1500 mg delivered once every 28 days.
  Other Names: (ABR-217620; NAP); (IMFINZI; MEDI4736)
  Arms: Dose Escalation naptumomab estafenatox 10 µg/kg and durvalumab; Dose Escalation naptumomab estafenatox 15 µg/kg and durvalumab; Dose Escalation naptumomab estafenatox 2 µg/kg and durvalumab; Dose Escalation naptumomab estafenatox 20 µg/kg and durvalumab; Dose Escalation naptumomab estafenatox 5 µg/kg and durvalumab

SUMMARY:
This Phase 1b is a dose escalation, MTD expansion and cohort expansions study to assess the safety and tolerability of a combination of NAP with durvalumab in subjects with selected advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This Phase 1b study was originally designed for patients with tumors reported to have a high probability of expressing the 5T4 antigen. An amended protocol extended the eligibility criteria of patients recruited to the maximum tolerated dose (MTD) cohort, to include colorectal cancer (CRC) and GE carcinomas.

Following the Dose Escalation part, antibodies binding to NAP have been shown to interfere with drug exposure, which makes it unlikely that patients could effectively receive more than 3 cycles of NAP. Obinutuzumab pretreatment was added to the combination of durvalumab and NAP given at the 2 highest safe dose levels of the combination of durvalumab and NAP in the dose-escalation part of this Phase 1b study (3 patients per dose level), and to the MTD expansion part that included several cohorts.

The combination of NAP/durvalumab combination will be further evaluated at the Recommended Phase 2 Dose (RP2D) established in the dose- escalation part, (10 µg/kg/dose), in an expansion cohort of subjects with advanced/metastatic carcinoma of the esophagus.

ELIGIBILITY:
Subjects must meet all of the following criteria to participate in this study:

1. Adult at least 18 years of age
2. For the Dose-escalation and MTD Expansion Cohorts: Histologically and/or cytologically confirmed solid tumor from the following list, that is metastatic/advanced, and for which no curative therapy exists:

   1. Pancreatic adenocarcinoma
   2. High-grade serous ovarian cancer
   3. Cervical squamous cell carcinoma
   4. Prostate cancer
   5. ER+/HER2- or triple-negative breast cancer
   6. NSCLC including driver mutation positive.
   7. Mesothelioma
   8. Renal cell carcinoma
   9. Bladder/urothelial cancer
   10. Head and neck squamous cell carcinoma
   11. Melanoma
   12. Hepatocellular carcinoma
   13. Endometrial cancer
   14. MTD Expansion Cohort only: 5T4-positive colorectal cancer and 5T4 positive GE cancer
3. For the Esophageal Expansion Cohort: Subjects must have histologically confirmed locally advanced or metastatic ESCC or AC of the esophagus or GEJ (Siewert type 1).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. All patients must provide signed informed consent prior to any study specific procedures that are not part of standard medical care.
6. In the MTD Expansion Cohort only, an archival or fresh biopsy will be acceptable at baseline. A second biopsy on Cycle 2 Day 4 is optional for patients who provided a fresh biopsy at baseline or have a tumor sample available from up to 3 months prior to study entry. Patients enrolled in the MTD expansion cohort after prior exposure to a CPI should have a baseline biopsy obtained after completion of the last prior CPI therapy.

   For the Esophageal Cohort Expansion: Subjects must have adequate tumor tissue (as defined in the laboratory manual) for biomarker analysis. If the archival tissue was taken > 1 year prior to screening into the trial, a fresh biopsy is required. Patients enrolled in Group 2 should have a baseline biopsy obtained after completion of the last prior CPI therapy. Bone samples, fine needle aspirates, brushings, cell pellets, and lavage are not acceptable samples.
7. Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 28 days prior to Cycle 1 Day 1 (first NAP treatment day)

   1. Dose-escalation part: patients do not need to have measurable disease by RECIST 1.1
   2. MTD Dose Expansion: patients must have measurable disease by iRECIST/RECIST 1.1. Previously irradiated lesions may be considered measurable if there has been demonstrated progression in these lesions.
   3. For the Esophageal Cohort Expansion: Patients must have measurable disease per iRECIST/RECIST version 1.1 by local investigator/ radiology assessment, unresectable based on documented opinion, or refusing surgery.
8. Previous therapy:

   a. Dose Escalation and MTD Expansion: i. All patients must have received at least 1 standard systemic cancer therapy for their tumor type and progressed following their most recent regimen. There is no limit to the number of prior cytotoxic regimens received.

   ii. Treatment-naïve patients will be eligible only if they refused standard treatment.

   iii. Patients with prior anti-PD-1, anti PD-L1, or anti-CTLA4 therapy are eligible if they have received such therapy for a minimum of 6 months and if they have documented progression of their disease on or off such therapy.

   b. Esophageal Cohort Expansion: i. Group 1 - no prior CPI: Subjects with only ESCC who may have received up to 1 prior chemotherapy as a line for metastatic disease or up to 2 prior chemotherapies if they also received neoadjuvant/adjuvant systemic therapy, but no prior CPI.

   If subjects received prior chemotherapy for metastatic disease, they should have documented radiographic or clinical progression.

   ii. Group 2 - prior CPI: Subjects with either ESCC or AC of the esophagus or GEJ (Siewert type 1) who must not have had more than 2 prior lines of therapy. Patients will be allowed to have up to 2 prior regimens for metastatic disease, or up to 3 prior therapies if they also received neoadjuvant/adjuvant systemic therapy.

   Subjects are eligible provided that they have received CPI therapy for at least 9 weeks, provided that they have documented progression of their disease on such therapy, and provided that the prior CPI was not discontinued for toxicity.

   No more than 1 prior CPI treatment is allowed (prior combination of anti-PD-[L]1 and anti-CTLA-4 is acceptable).

   Subjects with AC that is HER 2/neu negative.
9. Subjects with known, suspected, or documented parenchymal brain metastases, unless treated with surgery and/or radiation, with the subject neurologically stable and off pharmacologic doses of systemic glucocorticoids (equivalent to < 10 mg/day of prednisone); subjects with leptomeningeal metastases are not eligible. Subjects should have completed brain radiation at least 14 days before start of obinutuzumab treatment.
10. Prior treatment with chemotherapy or other systemic antineoplastic therapy within 21 days; prior experimental therapy within 21 days or 5 half-lives, whichever is shorter.
11. The use of immunosuppressive agents within 28 days of obinutuzumab administration including, but not limited to, cyclosporine, mycophenolate, azathioprine, methotrexate, adalimumab, infliximab, vedolizumab, tofacitinib, dupilumab, rituximab, etc. Pharmacologic doses of glucocorticoids defined as glucocorticoid equivalents of > 10 mg/day of prednisone (except when required for study medications or used prior to administration of radiographic contrast material in subjects with allergies) are not acceptable within 14 days of obinutuzumab administration. Subjects are permitted to receive topical, intranasal, inhalational, and intra ocular glucocorticoids.
12. Adequate hematologic and organ function:

    1. White blood cells (WBC) ≥ 3000/μL
    2. Absolute neutrophil count (ANC) ≥ 1500/μL
    3. Platelets ≥ 100,000/μL
    4. Hemoglobin ≥ 9 g/dL
    5. Serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance (CrCL) > 40 mL/sec by Cockcroft-Gault (using actual body weight)
    6. Aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) ≤ 2.5 × ULN (for patients with known liver involvement AST and ALT ≤ 5 × ULN); bilirubin ≤ 1.5 mg/dL (unless diagnosed with Gilbert's syndrome)
    7. International normalized ratio (INR) or prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. Subjects on anticoagulant therapy should be discussed with the Medical Monitor.
13. Patients must be willing and able to comply with scheduled visits, drug administration plan, hospitalization for treatment (if needed) and scheduled follow-up visits and examinations as outlined in the protocol, including procedures undertaken to perform fresh tumor biopsies if needed.
14. Must have a life expectancy of at least 3 months.
15. Negative pregnancy test (serum) for women of childbearing potential.
16. Female participants must be ≥ 1 year post-menopausal, surgically sterile, or using 1 highly effective form of birth control (a highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly.) Women of childbearing potential must agree to use 1 highly effective method of birth control. They should have been stable on their chosen method of birth control for a minimum of 3 months before entering the study until 90 days after the last dose of NAP + durvalumab combination therapy or durvalumab monotherapy. Non sterilized male partners of a female subject of childbearing potential must use a male condom plus spermicide throughout this period.
17. Male participants who intend to be sexually active with a female partner of childbearing potential must be surgically sterile or using an acceptable method of contraception from the time of Screening throughout the total duration of the study and until 90 days after the last dose of NAP + durvalumab combination therapy or durvalumab monotherapy to prevent pregnancy in a partner. Male participants must not donate or bank sperm during this same time period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Part A: Dose Escalation / MTD Expansion: The incidence and characteristics of adverse events, associated with ascending doses of NAP in combination with a set dose of durvalumab | From day 1 up to 90 days following last dose of study drug
  Number of participants with infusion reactions, Dose Limiting Toxicity (DLT) during the first cycle of treatment and/or, any adverse events graded as per NCI Common Toxicity Criteria (CTC).
Part A: Dose Escalation / MTD Expansion: The incidence and characteristics of adverse events, associated with ascending doses of NAP in combination with a set dose of durvalumab and following pretreatment with obinutuzumab. | From day -13 up to 90 days following last dose of study drug
  Number of participants with infusion reactions (e.g. fever, chills, hypotension, tachycardia etc.), occurrence of any Dose Limiting Toxicity (DLT) during the first cycle of treatment and/or , any clinically significant changes from baseline graded as per NCI Common Toxicity Criteria (CTC).
Part A: Dose Escalation / MTD Expansion: The RP2D either with or without obinutuzumab pretreatment | From day -13 up to 90 days following last dose of study drug
  based on the observed safety effects in the DE and MTD expansion cohorts.
Part B: Esophageal Cohort Expansion - ORR | 24 month
  The ORR by immune therapy-based Response Evaluation Criteria in Solid Tumours (iRECIST) of the combination of NAP with durvalumab in subjects with advanced/metastatic:
  1. ESCC without exposure to prior anti PD-1/PD-L1 therapy (Group 1), OR
  2. Squamous cell carcinoma or AC of the esophagus or GEJ who have received prior anti PD-1/PD-L1 therapy (Group 2).

SECONDARY OUTCOMES:
Part A: Dose Escalation / MTD Expansion: Disease parameters: ORR, DOR, PFS, OS | From date of initiation of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months post last patient in.
  Tumor assessment for ORR, DOR and PFS according to the iRECIST and conventional RECIST 1.1. OS will be based on death events.
Part A: Dose Escalation: Establish Recommended Phase 2 Dose (RP2D) | From Day 1 up to end of cycle 3 of dose escalation cohort without obinutuzumab
  RP2D will be determined based on the observed effects of the MTD.
Part A: Dose Escalation / MTD Expansion: Assessment of anti-NAP antibody levels and human anti-murine antibody (HAMA) levels at the beginning of each treatment cycle. | From start of treatment till end of cycle 3 in dose escalation and end of cycle 6 in MTD expansion (each cycle is 21 days).
  Blood levels of ADAs and HAMA
Part A: Dose Escalation / MTD Expansion: Assessment of NAP plasma levels at select time points | From start of treatment till end of cycle 3 in dose escalation and end of cycle 6 in MTD expansion (each cycle is 21 days).
  Pharmacokinetic calculations will be based on individual subject NAP plasma concentrations over time
Part B: Esophageal Cohort Expansion: ORR | 24 month
  1. The ORR by RECIST version 1.1 criteria, of the combination of NAP with durvalumab in subjects who are CPI naïve (ESCC; Group 1) and in subjects previously treated with a CPI (ESCC, AC; Group 2).
Part B: Esophageal Cohort Expansion: OS, PFS, DOR, rate & duration of disease control | 24 month
  2. To assess the following efficacy parameters in each group:
  1. OS, defined as time of enrolling on study (start of any study treatment) to death from whatever cause.
  2. PFS (by iRECIST and RECIST 1.1.), defined as the time of enrolling on study (start of any study treatment) to disease progression or death from whatever cause.
  3. DOR (by iRECIST and RECIST 1.1.) in subjects who achieve an objective response (CR or PR) defined as the time from first evidence of response to PD.
  4. Rate and duration of disease control (by iRECIST and RECIST 1.1.) in patients with CR, PR, or SD.
Part B: Esophageal Cohort Expansion: safety and tolerability | 24 month
  3. Assessment of the safety and tolerability of NAP/durvalumab combination:
  1. Safety will be measured by the incidence of treatment emergent adverse events (TEAEs), changes from baseline in vital signs, findings on physical examinations, ECGs, blood chemistry, complete blood count (CBC), urine and thyroid function laboratory tests, and graded per NCI CTCAE.
  2. Adverse events of special interest will include immune-based, tissue specific autoimmune conditions (e.g., colitis, pneumonitis).
  3. Tolerability will be measured by dose interruptions, dose reductions (NAP) and discontinuations due to drug-related AEs.
Part B: Esophageal Cohort Expansion: Assessment of NAP plasma levels at select time points and ADAs | 24 month
  4. Assessment of plasma levels of total NAP and ADAs (to be analyzed centrally at Labcorp).

CONTACTS AND LOCATIONS:
Overall Officials: Tal Hetzroni Kedem, Study Director — NeoTX Therapeutics Ltd.
Locations (9):
- India (5):
  - Shalby Hospital, Ahmedabad, Gujarat
  - National Cancer Institute, Jhajjar, Haryana
  - All India Institute of Medical Sciences, New Delhi, New Delhi
  - PMCH (Pacific Medical College & Hospital), Udaipur, Rajasthan
  - Basavatarakam Indo-American Cancer Hospital & Research Institute, Hyderabad, Telangana
- Israel (4):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No